CLINICAL TRIAL: NCT04825509
Title: Ultrasound-Assessed Diaphragmatic Dysfunction as a Predictor of Weaning Outcome in Mechanically Ventilated Patients With Sepsis in Intensive Care Unit
Brief Title: Ultrasound-Assessed Diaphragmatic Dysfunction as a Predictor of Weaning Outcome
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Saad, Dr, Ain Shams University
Other Study IDs: Diaphragm Ultrasound
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Weaning Failure; Sepsis
Keywords: Diaphragm ultrasound; Weaning predictor
MeSH Terms: conditions — Sepsis | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Successful weaning group: Patients will be in this group according to primary outcome, if they will succeed spontaneous breathing trial for 120 minutes and will be extubated successfully without need for invasive or non-invasive ventilation for 48 hours
  Interventions: Device: Ultrasound
- Weaning failure group: Patients will be in this group according to primary outcome, if they will fail spontaneous breathing trial or extubation within 48 hours
  Weaning failure will be considered if:
  * Patients will need MV during spontaneous breathing trial within 120 minutes, or
  * patients will need invasive or non-invasive ventilation within 48 hours
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Diaphragm ultrasound will be done while patient is supine on T-piece during SBT 30 minutes after disconnecting mechanical ventilation. The measurements will be done by placing the transducer in the eighth or ninth intercostal space, between the anterior axillary and the mid-axillary lines.
  Diaphragmatic excursion (DE) will be measured in M-mode using a 1- to 5- Megahertz (MHz) ultrasound curved transducer during maximal breathing. The amplitude of diaphragmatic excursion will be measured as the point of maximal height of the diaphragm to the base line.
  Diaphragmatic thickness (DT) will be measured at both end of maximal inspiration and end of maximal expiration using a high frequency 7-11 MHz ultrasound linear transducer in M-mode. The diaphragm thickness will be measured from the middle of the pleural line to the middle of the peritoneal line.

SUMMARY:
This study aims to assess whether the degree of diaphragm excursion and diaphragm thickening measured by ultrasound during a weaning trial may be used to predict successful weaning from mechanical ventilation in patients with sepsis in intensive care unit

DETAILED DESCRIPTION:
After being informed about the study and giving written informed consent, Intubated and mechanically ventilated patients with sepsis on admission and fulfilling criteria of weaning from mechanical ventilation (MV), will undergo diaphragm ultrasound during spontaneous breathing trial on T-piece. We will measure diaphragm excursion (DE), diaphragm thickness (DT) and calculate diaphragm thickness fraction (DTF):

DT during inspiration - DT during expiration / DT during expiration

According to weaning outcome, patients will be divided into 2 groups:

* Successful weaning group
* Weaning failure group

By statistical analysis we will define the cut off value and area under curve (AUC) for DE and DTF and we can confirm if DE and DTF using ultrasound can be used as predictors for weaning from MV or not

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, aging 18 - 60 years after written informed consent
* Patients with sepsis on admission according to the new sepsis definition in 2016 (life-threatening organ dysfunction due to a dysregulated host response to infection)
* Hemodynamically stable without or with low dose support
* Patients on mechanical ventilation for at least 48 hours and not more than 1 week
* Patients ready for start of weaning protocol, fully conscious, on continuous positive airway pressure (CPAP) mode with positive end expiratory pressure (PEEP) 3-5 Centimetre water (CmH2O), Pr. Supp. <15 CmH2O, Fio2 less than 60%, Respiratory rate less than 35 breath/min, partial oxygen pressure (PO2)/FIO2 >200, Rapid Shallow Breathing Index (RSBI) is less than 105

Exclusion Criteria:

* Patients aged less than 18 years or more than 60 years old
* Patients in septic shock, hemodynamically unstable or on high dose support
* Patients on mechanical ventilation for more than 1 week or less than 48 hours
* Patients not ready for start of weaning from mechanical ventilation
* Patients with neuromuscular disorders
* Pregnant females in the second and third trimester, patients with tense ascites or morbidly obese with body mass index more than 40 kg/m2

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients will be intubated (for 2 - 7 days) and ready for weaning process. They will undergo diaphragmatic ultrasound on spontaneous breathing pattern on T-piece connected to 8L/min O2 with subsequent outcome either successful weaning or failed weaning
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-04-18 (Actual); Primary Completion 2021-10-17 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Successful extubation | from start of SBT till 48 hours after extubation
  extubation success or failure will depend on patient needs to MV during spontaneous breathing trial (SBT), or invasive or non-invasive ventilation within 48 hours after extubation according to: respiratory rate>35/min, increased work of breathing, O2 saturation <90% with fraction of inspired oxygen (FIO2)>50%, new arrhythmias, increased heart rate>20% or more than 140b/min, drop of 20 millimetre mercury (mmHg) or rise of 30 mmHg systolic blood pressure, increased systolic blood pressure >180 mmHg in normotensive patient, change of 10 mmHg diastolic blood pressure and deterioration of blood gases value

SECONDARY OUTCOMES:
need for tracheostomy | From start of SBT for 21 days
  We will check patient need for tracheostomy since start of weaning process for 21 days and the indication for tracheostomy, if due to prolonged intubation or other causes

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Saad, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual patient data (IPD) that underlie the results reported in this article after deidentification (texts, tables, figures and appendices) will be available only for investigators whose purposed use of the data has been approved by an independent review committee identified for this purpose

REFERENCES:
- [Background] Llamas-Alvarez AM, Tenza-Lozano EM, Latour-Perez J. Diaphragm and Lung Ultrasound to Predict Weaning Outcome: Systematic Review and Meta-Analysis. Chest. 2017 Dec;152(6):1140-1150. doi: 10.1016/j.chest.2017.08.028. Epub 2017 Aug 31. PMID 28864053
- [Background] DiNino E, Gartman EJ, Sethi JM, McCool FD. Diaphragm ultrasound as a predictor of successful extubation from mechanical ventilation. Thorax. 2014 May;69(5):423-7. doi: 10.1136/thoraxjnl-2013-204111. Epub 2013 Dec 23. PMID 24365607
- [Background] Kilaru D, Panebianco N, Baston C. Diaphragm Ultrasound in Weaning From Mechanical Ventilation. Chest. 2021 Mar;159(3):1166-1172. doi: 10.1016/j.chest.2020.12.003. Epub 2020 Dec 10. PMID 33309837